CLINICAL TRIAL: NCT04460352
Title: NEoadjuvant Chemoradiotherapy for Esophageal Squamous Cell Carcinoma Versus Definitive Chemoradiotherapy With Salvage Surgery as Needed (NEEDS Trial)
Brief Title: Chemoradiotherapy Followed by Planned Surgery or by Surveillance and Surgery Only When Needed for Oesophageal Cancer
Acronym: NEEDS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: University of Leipzig (Other); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Magnus Nilsson, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEEDS
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Neoadjuvant chemoradiotherapy; Definitive chemoradiotherapy with salvage surgery as needed
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Neoadjuvant Therapy; CP protocol; Esophagectomy; TP protocol; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: NEEDS is a pragmatic open-label, randomised, controlled, phase III, multicenter trial with non-inferiority design with regard to the three co-primary endpoints i) Overall survival and superiority for the experimental intervention definitive chemoradiotherapy; ii) Global health related quality of life (HRQOL) one year after randomisation; iii) Eating restictions one year after randomisation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (A) (Active Comparator): Neoadjuvant chemoradiotherapy followed by esophagectomy.
  Radiotherapy: 1.8 Gy fractions 5 days per week in 23 fractions to a total dose of 41.4 Gy.
  Chemotherapy: Carboplatin AUC 2 + Paclitaxel 50mg/m2 weekly x 5 (day 1, 8, 15, 22, 29), starting on the first day of radiotherapy.
  Esophagectomy: Within 8 weeks of termination of chemoradiotherapy,
  Interventions: Radiation: Neoadjuvant radiotherapy (arm A); Drug: Carboplatin, paclitaxel; Procedure: Esophagectomy
- Experimental arm (B) (Experimental): Definitive chemoradiotherapy followed by surveillance, and esophagectomy only in case of residual or recurrent locoregional cancer.
  Radiotherapy: Two alternative schemes:
  1. 1.8 Gy fractions five days per week in 28 fractions to a total dose of 50.4 Gy.
  2. 2.0 Gy fractions five days per week in 25 fractions to a total dose of 50 Gy.
  Chemotherapy: Three alternative regimens:
  1. Platin-Taxane Regimen: Carboplatin AUC 2 + Paclitaxel 50mg/m2 on day 1 weekly during the full course of radiotherapy.
  2a. Platinum-Fluoropyrimidine Regimen: Cisplatin 75mg/m2 weeks 1 and 5 + 5-fluorouracil 1000 mg/m2/day by continuous infusion weeks 1 and 5.
  2b. FOLFOX: Oxaliplatin 85 mg/m2, calcium folinate 200 mg/m2 and 5-fluorouracil 400 mg/m2 weeks 1, 3 and 5 + 5-fluorouracil 800 mg/m2 by continuous infusion weeks 1, 3 and 5.
  Interventions: Radiation: Neoadjuvant radiotherapy (arm B); Drug: Carboplatin, paclitaxel; Drug: Cisplatin, paclitaxel; Drug: Oxaliplatin, calcium folinate, 5-fluorouracil; Procedure: Esophagectomy

INTERVENTIONS:
Radiation: Neoadjuvant radiotherapy (arm A) — 1.8 Gy fractions 5 days per week in 23 fractions to a total dose of 41.4 Gy.
  Arms: Control arm (A)
Drug: Carboplatin, paclitaxel — Carboplatin AUC 2 + Paclitaxel 50mg/m2 weekly x 5 (day 1, 8, 15, 22, 29), starting same day as radiotherapy
  Other Names: Neoadjuvant chemotherapy
  Arms: Control arm (A)
Procedure: Esophagectomy — Esophagectomy performed within 8 weeks after termination of chemoradiotherapy
  Arms: Control arm (A)
Radiation: Neoadjuvant radiotherapy (arm B) — Two alternative schemes:
  1. 1.8 Gy fractions five days per week in 28 fractions to a total dose of 50.4 Gy.
  2. 2.0 Gy fractions five days per week in 25 fractions to a total dose of 50 Gy.
  Arms: Experimental arm (B)
Drug: Carboplatin, paclitaxel — Carboplatin AUC 2 + Paclitaxel 50mg/m2 on day 1 weekly during the full course of radiotherapy (5 weeks or 6 weeks, depending on the radiotherapy regimen used).
  Other Names: Neoadjuvant Platin-Taxane Regimen (alternative 1)
  Arms: Experimental arm (B)
Drug: Cisplatin, paclitaxel — Cisplatin 75mg/m2 on the first day of weeks 1 and 5 + 5-fluorouracil 1000 mg/m2/day by continuous infusion on the first four days of weeks 1 and 5.
  Other Names: Platinum-Fluoropyrimidine Regimens (alternative 2a)
  Arms: Experimental arm (B)
Drug: Oxaliplatin, calcium folinate, 5-fluorouracil — FOLFOX: Oxaliplatin 85 mg/m2, calcium folinate 200 mg/m2 and 5-fluorouracil 400 mg/m2 on the first days of weeks 1, 3 and 5 + 5-fluorouracil 800 mg/m2 by continuous infusion on the first two days of weeks 1, 3 and 5.
  Other Names: Platinum-Fluoropyrimidine Regimens (alternative 2b)
  Arms: Experimental arm (B)
Procedure: Esophagectomy — Esophagectomy only in case of residual or recurrent locoregional cancer.
  Arms: Experimental arm (B)

SUMMARY:
NEEDS is a pragmatic open-label, randomised, controlled, phase III, multicenter trial with non-inferiority design with regard to the first co-primary endpoint overall survival and superiority for the experimental intervention definitive chemoradiotherapy. A second co-primary endpoint is global health related quality of life (HRQOL) one year after randomisation. A third co-primary endpoint is eating restictions one year after randomisation.

The aim is to compare outcomes after neoadjuvant chemoradiotherapy with subsequent esophagectomy to definitive chemoradiotherapy with surveillance and salvage esophagectomy as needed in patients with resectable locally advanced squamous cell carcinoma (SCC) of the esophagus, with the aim to provide generalisable guidance for future clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed SCC of the esophagus in locally advanced stages cT1 N+ or cT2-4a any N, M0, according to current (8th) version of of the AJCC TNM classification.
* Technically resectable disease according to the local multidisciplinary team conference (MDT)/tumor board.
* Performance status ECOG 0-1.
* Adequate organ function.
* Women of childbearing potential (WOCBP*) must have a negative serum or urine pregnancy test.
* Patients of childbearing/reproductive potential should use highly effective method of birth control measures during the study treatment period and for at least five months after the last study treatment.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP/GDPR and national/local regulations.

Exclusion Criteria:

* M1 according to current (8th) version of of the AJCC TNM classification.
* cT4b according to current (8th) version of of the AJCC TNM classification.
* Primary tumor not resectable without laryngectomy.
* Impaired renal, hepatic, cardiac, pulmonary or endocrine status that compromises the eligibility of the patient for multimodality treatment with chemoradiotherapy followed by esophagectomy.
* Subjects not considered likely to tolerate multimodality treatment with chemoradiotherapy followed by esophagectomy.
* Subjects with previous malignancies are excluded unless a complete remission or complete resection was achieved at least 5 years prior to study entry.
* Prior or concomitant treatment with radiotherapy or chemoradiotherapy with potential overlap of radiotherapy fields.
* Known uncontrollable hypersensitivity to the components of the chemotherapeutic agents used in the trial regimens.
* Inability to fully understand and digest study patient information or to comply with study instructions due to language difficulty or cognitive failure such as dementia or severe psychiatric disorder.

(Criteria slightly shortened)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years after randomisation
  When 398 events have occurred
Global Health-related quality of life (HRQOL) | 1 year after randomisation
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-C30, version 3.0 (EORTC QLQ-C30). The two items assessing global health and overall quality of life are responded to in seven categories ranging from 1 (very poor) to 7 (excellent).
Eating restrictions | 1 year after randomisation
  EORTC QLQ-OG25 instrument. This instrument consists of 25 items covering upper gastric symptoms or problems in four categories ranging from 1 (Not at all) to 4 (Very much).

SECONDARY OUTCOMES:
Health related quality of life of Cancer patients | At randomisation but before start of treatment and thereafter 6, 12, 24, 36 and 60 months after randomisation
  EORTC HRQOL Questionnaire QLQ-C30 version 3.0, 28 items ranging from 1 (no problems at all) to 4 (very much) and two items assessing global health and overall quality of life are responded to in seven categories ranging from 1 (very poor) to 7 (excellent).
Health related quality of life, oesophageal specific. | At randomisation but before start of treatment and thereafter 6, 12, 24, 36 and 60 months after randomisation
  EORTC HRQOL gastresophageal-specific questionnaire EORTC QLQ-OG25. 25 items assessing symptoms or problems are responded to in four categories ranging from 1 (no problems) to 4 (very much).
Health related quality of life, general health | At randomisation but before start of treatment and thereafter 6, 12, 24, 36 and 60 months after randomisation
  The EuroQoL Group's EQ-5D-5L questionnaire consisting of five dimensions ranging from No problems to Extreme problems or Unable to care.
Event-free survival | 5 years after randomisation
  Time to relapse, initiation of any anti-tumor therapy beyond the study treatments (salvage surgery is considered a study treatment in the dCRT arm), or death, whichever comes first.
Loco-regional and distant relapse rates | 5 years after randomisation
  Including the relation of relapse location to the radiation field
Histopathological response according to Mandard in operated patients | 5 years after randomisation
  ypTNM including total and metastatic lymph node count, tumor free resection margins, R0
Health economy | At baseline and 6, 12, 24, 36 and 60 months after randomisation
  Assessed including patient-level medical resource use and societal costs due to sick-leave and other non-medical costs. Quality-adjusted life years (QALYs) will be calculated using EQ-5D
Surgical complications | After surgery in operated patients, up to 5 years after randomisation
  According to the Esophagectomy Complications Consensus Group (ECCG) and classified according to Clavien-Dindo
Treatment-related adverse events and toxicity | Up to 5 years after randomisation
  NCI-CTCAE Criteria version 5.0
Nutritional outcomes - weight | Up to 5 years after randomisation
  Weight development. Weight (in kg) will be measured at all visits.
Nutritional outcomes - dysphagia | Up to 5 years after randomisation
  Dysphagia will be evaluated at all visits according to the CTC adverse event scale, grading from 0 (no problems) to 4 (worst problems).
Gender stratified analyses of all endpoints | Up to 5 years after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Nilsson, MD, PhD, Study Chair — Karolinska University Hospital; Florian Lordick, MD, PhD, Study Chair — Leipzig University Medical Center
Locations (12):
- McGill University Health Centre, Montreal, Quebec, Canada
- Cancer Clinical Trials Unit (CCTU) at St. James's Hospital, Dublin, Dublin, Ireland
- Norway (3):
  - Oslo universitetssykehus, Oslo
  - Universitetssykehuset Nord-Norge, Tromsø
  - St Olavs Hospital, Trondheim
- Sweden (6):
  - Linköpings universitetssjukhus, Linköping
  - Skånes universitetssjukhus, Lund
  - Örebro universitetssjukhus, Örebro
  - Karolinska University Hospital, Stockholm
  - Norrlands universitetssjukhus, Umeå
  - Akademiska sjukhuset, Uppsala
- Chang Gung Memorial Hospital, Linkou District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson M, Olafsdottir H, Alexandersson von Dobeln G, Villegas F, Gagliardi G, Hellstrom M, Wang QL, Johansson H, Gebski V, Hedberg J, Klevebro F, Markar S, Smyth E, Lagergren P, Al-Haidari G, Rekstad LC, Aahlin EK, Wallner B, Edholm D, Johansson J, Szabo E, Reynolds JV, Pramesh CS, Mummudi N, Joshi A, Ferri L, Wong RK, O'Callaghan C, Lukovic J, Chan KK, Leong T, Barbour A, Smithers M, Li Y, Kang X, Kong FM, Chao YK, Crosby T, Bruns C, van Laarhoven H, van Berge Henegouwen M, van Hillegersberg R, Rosati R, Piessen G, de Manzoni G, Lordick F. Neoadjuvant Chemoradiotherapy and Surgery for Esophageal Squamous Cell Carcinoma Versus Definitive Chemoradiotherapy With Salvage Surgery as Needed: The Study Protocol for the Randomized Controlled NEEDS Trial. Front Oncol. 2022 Jul 13;12:917961. doi: 10.3389/fonc.2022.917961. eCollection 2022. PMID 35912196